CLINICAL TRIAL: NCT06319898
Title: Relaxing Environment to Lower Anxiety During Onabotulinum Toxin Chemodenervation of the Bladder: RELAX Trial
Brief Title: Relaxing Environment to Lower Anxiety During Onabotulinum Toxin Chemodenervation of the Bladder
Acronym: RELAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00110787
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Results first posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-02

CONDITIONS: Anxiety; Pain; Burnout, Professional
Keywords: aromatherapy; bladder botox; anxiety; lavender
MeSH Terms: conditions — Anxiety Disorders; Pain; Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lavender aromatherapy sticker (Experimental): Lavender aromatherapy sticker on patient Calming music from Sirius station 68 (Spa) playing via overhead speakers Overhead lights off, two lanterns lit to provide dim lighting Avoid stirrup use
  Interventions: Behavioral: Lavender aromatherapy sticker
- Control - no Intervention (No Intervention): Non-aromatic (placebo) sticker on patient No music playing Overhead lights on Stirrups used
- Procedure Team Intervention - relaxing environment (Experimental): lavender aromatherapy, calming music, and dim lighting - Members of the procedure team - participation in this research will involve a 3 question initial questionnaire survey to assess demographics and prior experience with aromatherapy and pre- and post-clinic survey on the days you participate in bladder Botox procedures.
  Interventions: Behavioral: Lavender aromatherapy sticker
- Procedure Team Control - no Intervention (No Intervention): Members of the procedure team - participation in this research will involve a 3 question initial questionnaire survey to assess demographics and prior experience with aromatherapy and pre- and post-clinic survey on the days you participate in bladder Botox procedures.

INTERVENTIONS:
Behavioral: Lavender aromatherapy sticker — Lavender aromatherapy during procedure, music and dim lighting
  Other Names: music and dim lighting
  Arms: Lavender aromatherapy sticker; Procedure Team Intervention - relaxing environment

SUMMARY:
Chemodenervation of the bladder with onabotulinum toxin A is an effective treatment option for patients with refractory urgency urinary incontinence (UUI). It is often performed as an office-based procedure under local anesthesia. Alternatively, it can be performed in the operating room under general anesthesia. The ability to receive intra-detrusor chemodenervation in the office allows patients to avoid the risks associated with general anesthesia and is significantly more cost effective. The procedure, however, is painful and can be anxiety provoking for patients; especially given that patients typically return every six to nine months for repeat injections. Relaxation and distraction techniques are one way to ease patients' anxiety before an office-based procedure. While we do not know exactly how anxiety provoking office bladder chemodenervation is for patients, we do know that anxiety disorders are highly prevalent in women with overactive bladder as a population.

The purpose of this study is to investigate whether women with Urge urinary incontinence (UUI) who receive office intra-detrusor chemodenervation injections performed in a relaxing environment of lavender aromatherapy, calming music, dim lighting, and modest positioning (Relaxing Environment Package) will have decreased anxiety and pain as well as increased post-procedure satisfaction compared to patients who receive chemodenervation in a typical office environment. Also investigate whether exposure to the relaxing environment impacts the well-being of staff involved in these procedures. This study design is a randomized control trial. Women scheduled for office intra-detrusor chemodenervation at Atrium Health women's Care Urogynecology & Pelvic Surgery - Mercy clinic will be invited to participate. Participants will be randomized to the relaxing environment package or the placebo group after informed consent is obtained and immediately before undergoing intra-detrusor chemodenervation. The participants will complete the pre-procedure visual analog scale (VAS) for anxiety and a VAS for pain at baseline.

DETAILED DESCRIPTION:
Aside from randomization to relaxing environment package versus placebo, no procedures will be performed for study purposes that would not be normally performed in the clinical evaluation.

Women scheduled for office intra-detrusor chemodenervation at Atrium Health women's Care Urogynecology & Pelvic Surgery - Mercy, Charlotte North Carolina, will be invited to participate. Participants who meet inclusion criteria will be randomized to the relaxing environment package or the placebo group after informed consent is obtained and immediately before undergoing intra-detrusor chemodenervation. Randomization of weeks rather than individual participants was selected to minimize impact to clinic flow. A permuted block randomization scheme will be used to assign weeks in a 1:1 ratio to intervention or control. After obtaining informed consent, all participants will fill out a baseline pre-procedural visual analog scale (VAS) for anxiety and a VAS for pain. Anxiety will be assessed using a visual analog scale (VAS)

If the week is randomized to a Relaxing Environment Package week, the patient, procedure staff, and MD will enter the procedure room and receive a lavender aromatherapy sticker to be worn on their lapels. Calming music from Sirius station 68 (Spa) will be playing softly in the background via overhead speakers. If the patient had planned to listen to their own music during the procedure, this will be permitted. The overhead lights will then be turned off, and two lanterns lit to provide dim lighting. Stirrups will be avoided if possible, during the preparation and procedure.

If the week is randomized to Typical Office Environment, the patient, procedure staff, and MD will enter the procedure room and receive a non-aromatic (placebo) sticker to be worn on their lapels. No music will be playing, and all of the lights will be on as is typical in our practice. The lights may then be adjusted during cystoscopy per provider preference for adequate visualization.

All patients will receive routine preprocedural antibiotic prophylaxis, sterile urethral preparation with betadine or chlorhexidine, and 60cc viscous intravesical 1% lidocaine. After sitting in the environment for at least 10 minutes while the local anesthetic takes effect, participants will fill out a 2nd VAS for anxiety. The standard bladder chemodenervation procedure will be performed, and any patient requested modifications to the protocol will be recorded. After the procedure and once participants are dressed, they will fill out a 2nd VAS for pain and a VAS for procedure satisfaction. The VAS for patient satisfaction is a validated scale ranging from 0-100mm.

The procedure staff and MD will fill out the Burnout Battery visual analog scale for healthcare worker burnout at the start of the day before seeing any patients and again at the end of the day after seeing their last patient. This tool was created to assess the working energy states of healthcare providers and is correlated with the Maslach Burnout Inventory which is a validated 22 question survey regarding workplace burnout. They will also record how many chemodenervation procedures they participated in that day.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant females
* Age 18 years and older
* English as a primary language
* Scheduled for office intra-detrusor chemodenervation for diagnosis of Over-Active Bladder (OAB)/ Urinary Urgency (UU)/ Urged Urinary Incontinence (UUI)
* Baseline visual analog scale for anxiety ≥12mm

Exclusion Criteria:

* Allergy to lavender oil
* Contraindication to intra-detrusor chemodenervation (active Urinary Tract Infection)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 113 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Tarr, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Procedure Team Intervention - Relaxing Environment: Lavender aromatherapy, calming music and dim lighting
- Procedure Team - no Intervention: No intervention in Procedure Room
Period: Overall Study
Arm/Group | Lavender Aromatherapy Sticker | Control - no Intervention | Procedure Team Intervention - Relaxing Environment | Procedure Team - no Intervention
Started | 42 | 47 | 10 | 11
Completed | 40 | 40 | 10 | 11
Not Completed | 2 | 7 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Procedure Team Intervention - Relaxing Environment: Lavender aromatherapy Calming music Overhead lights off
- Procedure Team - no Intervention: Non-aromatic No music playing Overhead lights on
- Total: Total of all reporting groups
Arm/Group | Lavender Aromatherapy Sticker | Control - no Intervention | Procedure Team Intervention - Relaxing Environment | Procedure Team - no Intervention | Total
Number analyzed (Participants) | 40 | 40 | 10 | 11 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] — This measurement was not collected for the Procedure Team Members Population: This measurement was not collected on Procedure Team Intervention - Relaxing Environment and Procedure Team - no Intervention Groups
  years
    number analyzed (Participants) | 40 | 40 | 0 | 0 | 80
    (all) | 72.4 (11.6) | 69.1 (13.1) |  |  | 70.7 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 9 | 10 | 99
  Male | 0 | 0 | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: This measurement was not collected on Procedure Team Intervention - Relaxing Environment and Procedure Team - no Intervention Groups
  Participants
    number analyzed (Participants) | 40 | 40 | 0 | 0 | 80
    Hispanic or Latino | 1 | 0 |  |  | 1
    Not Hispanic or Latino | 38 | 40 |  |  | 78
    Unknown or Not Reported | 1 | 0 |  |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: This measurement was not collected on Procedure Team Intervention - Relaxing Environment and Procedure Team - no Intervention Groups
  Participants
    number analyzed (Participants) | 40 | 40 | 0 | 0 | 80
    American Indian or Alaska Native | 0 | 0 |  |  | 0
    Asian | 0 | 0 |  |  | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
    Black or African American | 4 | 7 |  |  | 11
    White | 35 | 33 |  |  | 68
    More than one race | 1 | 0 |  |  | 1
    Unknown or Not Reported | 0 | 0 |  |  | 0
Tobacco use [Count of Participants; unit: Participants] — Population: This measurement was not collected on Procedure Team Intervention - Relaxing Environment and Procedure Team - no Intervention Groups
  Participants
    Never smoker: number analyzed (Participants) | 40 | 40 | 0 | 0 | 80
    Never smoker | 28 | 23 | 0 | 0 | 51
    Former smoker: number analyzed (Participants) | 40 | 40 | 0 | 0 | 80
    Former smoker | 12 | 16 | 0 | 0 | 28
    Current smoker: number analyzed (Participants) | 40 | 40 | 0 | 0 | 80
    Current smoker | 0 | 1 | 0 | 0 | 1
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — Population: This measurement was not collected on Procedure Team Intervention - Relaxing Environment and Procedure Team - no Intervention Groups
  kg/m^2
    number analyzed (Participants) | 40 | 40 | 0 | 0 | 80
    (all) | 29.6 (6.7) | 30.9 (7.6) |  |  | 30.2 (7.1)
First-time bladder chemodenervation experience [Count of Participants; unit: Participants] — We documented if it was the patient's first time having the bladder chemodenervation procedure performed as this might impact their anxiety level compared to a patient who has experienced the procedure before. This measurement was not collected on Procedure Team Intervention - Relaxing Environment and Procedure Team - no Intervention Groups Population: This measurement was not collected on Procedure Team Members
  Participants
    yes: number analyzed (Participants) | 40 | 40 | 0 | 0 | 80
    yes | 9 | 8 | 0 | 0 | 17
    no: number analyzed (Participants) | 40 | 40 | 0 | 0 | 80
    no | 31 | 32 | 0 | 0 | 63
Anxiety diagnosis [Count of Participants; unit: Participants] — We recorded if patients had a documented anxiety diagnosis. Population: This measurement was not collected on Procedure Team Intervention - Relaxing Environment and Procedure Team - no Intervention Groups
  Participants
    yes: number analyzed (Participants) | 40 | 40 | 0 | 0 | 80
    yes | 7 | 10 | 0 | 0 | 17
    no: number analyzed (Participants) | 40 | 40 | 0 | 0 | 80
    no | 33 | 30 | 0 | 0 | 63
Pain medication use [Count of Participants; unit: Participants] — We recorded if pain medications were used in the last 24 hours prior to the procedure. Population: This measurement was not collected on Procedure Team Intervention - Relaxing Environment and Procedure Team - no Intervention Groups
  Participants
    yes: number analyzed (Participants) | 40 | 40 | 0 | 0 | 80
    yes | 10 | 13 | 0 | 0 | 23
    no: number analyzed (Participants) | 40 | 40 | 0 | 0 | 80
    no | 30 | 27 | 0 | 0 | 57
Insurance type [Count of Participants; unit: Participants] — Population: This measurement was not collected on Procedure Team Members
  Participants
    Private: number analyzed (Participants) | 40 | 40 | 0 | 0 | 80
    Private | 7 | 9 | 0 | 0 | 16
    Medicare: number analyzed (Participants) | 40 | 40 | 0 | 0 | 80
    Medicare | 31 | 29 | 0 | 0 | 60
    Medicaid: number analyzed (Participants) | 40 | 40 | 0 | 0 | 80
    Medicaid | 2 | 2 | 0 | 0 | 4
Aromatherapy use [Count of Participants; unit: Participants] — We recorded if patients had used aromatherapy in the past 6 months to help understand their familiarity with aromatherapy. Population: This measurement was not collected on Procedure Team Members
  Participants
    yes | 11 | 17 | 4 | 3 | 35
    no | 29 | 23 | 6 | 8 | 66
Years of Experience in current role [Mean (Standard Deviation); unit: years] — Population: This measurement was not collected for the Subjects acquiring Procedure
  years
    number analyzed (Participants) | 0 | 0 | 10 | 11 | 21
    (all) |  |  | 7.53 (9.24) | 10.41 (10.3) | 9.94 (9.98)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Visual Analog Scale (VAS) Anxiety Scores
Description: The VAS for anxiety is a validated scale that ranges from 0-100mm. 0mm is equivalent to "no anxiety" and is located on the left. 100mm is equivalent to "extremely anxious" and is located on the right. The minimum clinically important difference for VAS anxiety is a change of 12mm on a 100mm scale.
Time Frame: Baseline to Minute 30
Population: This Measurement was not collected from Procedure Team Members
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Procedure Team Intervention - Relaxing Environment: Lavender aromatherapy, calming music, and dim lighting
- Procedure Team Control - no Intervention: No aromatherapy or music - lights were on
Arm/Group | Lavender Aromatherapy Sticker | Control - no Intervention | Procedure Team Intervention - Relaxing Environment | Procedure Team Control - no Intervention
Number analyzed (Participants) | 40 | 40 | 0 | 0
mm | -13.8 (18.1) | -4.7 (14.7) |  |

2. Secondary Outcome: Mean Change in Visual Analog Scale (VAS) Pain During the Chemodenervation Procedure
Description: Pain during the chemodenervation procedure will be assessed using a visual analog scale for pain. The VAS for pain is a validated scale that ranges from 0-100mm12. 0mm is equivalent to "no pain" and is located on the left. 100mm is equivalent to "worst possible pain" and is located on the right. Subjects are asked to circle a number on the scale that corresponds to their level of pain during the procedure. Baseline scores will be collected on the day of the procedure in the research office after obtaining consent. Patients will then be asked to circle the pain scores that corresponded to the pain experienced during the procedure. This will be collected by study staff after the procedure once the patient is dressed.
Time Frame: Baseline to post-procedure up to 2 hours
Population: This measurement was not collected on Procedure Team Members
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Lavender Aromatherapy Sticker | Control - no Intervention | Procedure Team Intervention - Relaxing Environment | Procedure Team Control - no Intervention
Number analyzed (Participants) | 40 | 40 | 0 | 0
mm | 0.0 (23.4) | 3.7 (31.5) |  |

3. Secondary Outcome: Procedure Staff Burnout Scores - Burnout Battery Visual Analog Scale for Healthcare Worker Burnout
Description: Determine if the Relaxing Environment Package decreases procedure staff burnout based on Burnout Battery visual analog scale for healthcare worker burnout. This tool was created to assess the working energy states of healthcare providers and is correlated with the Maslach Burnout Inventory which is a validated 22 question survey regarding workplace burnout14. The clinic staff assigned to chemodenervation procedures as well as the physician performing the procedure will fill out the Burnout Battery VAS at the beginning and end of the clinic day. Providers are asked to circle the battery that represents their current energy level.
Time Frame: Baseline to post-procedure up to 2 hours
Population: This measurement was only collected for Procedure Team Members
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Procedure Team - no Intervention: No intervention in Procedure Room - no aromatherapy or music - lights were on
Arm/Group | Lavender Aromatherapy Sticker | Control - no Intervention | Procedure Team Intervention - Relaxing Environment | Procedure Team - no Intervention
Number analyzed (Participants) | 0 | 0 | 10 | 11
mm |  |  | -1.73 (1.78) | 1.31 (1.53)

4. Secondary Outcome: Patient Satisfaction With Their Procedure Experience Scores
Description: Patient satisfaction with their procedure experience will be assessed using a visual analog scale for patient satisfaction. The VAS for patient satisfaction is a validated scale ranging from 0-100mm. 0mm is equivalent to "no satisfaction" and 100mm is equivalent to "extreme satisfaction". Subjects are asked to circle a number that corresponds to their level of satisfaction with their procedure experience.
Time Frame: post procedure up to 2 hours
Population: This Measurement was not collected from Procedure Team Members
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Procedure Team Intervention - Relaxing Environment: lavender aromatherapy and music with dim lighting
Arm/Group | Lavender Aromatherapy Sticker | Control - no Intervention | Procedure Team Intervention - Relaxing Environment | Procedure Team Control - no Intervention
Number analyzed (Participants) | 40 | 40 | 0 | 0
mm | 91.4 (16.5) | 89.3 (19.0) |  |

ADVERSE EVENTS:
Time Frame: Hour 2
Groups:
- Control - no Intervention: Non-aromatic (placebo) sticker on patient No music playing Lavender aromatherapy sticker on patient Calming music from Sirius station 68 (Spa) playing via overhead speakers Overhead lights on Stirrups used
- Procedure Team Control - no Intervention: no aromatherapy or music - Overhead lights on
Arm/Group | Lavender Aromatherapy Sticker | Control - no Intervention | Procedure Team Intervention - Relaxing Environment | Procedure Team Control - no Intervention
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT06319898/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT06319898/ICF_001.pdf